CLINICAL TRIAL: NCT05098067
Title: Trial of Capsaicin Cream as an Adjunctive Therapy for Nausea and Vomiting of Pregnancy: A Pilot Investigation
Brief Title: Capsaicin Cream as an Adjunctive Therapy for Nausea and Vomiting of Pregnancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1763191-1
Record Dates: First submitted 2021-10-20; First posted 2021-10-28 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Hyperemesis Gravidarum; Nausea Gravidarum; Vomiting of Pregnancy
Keywords: capsaicin; nausea; vomiting; pregnancy; hyperemesis gravidarum
MeSH Terms: conditions — Hyperemesis Gravidarum; Nausea; Vomiting | interventions — Metoclopramide; Ondansetron; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group (Experimental): Participants will receive IV fluid bolus of 1000cc of lactated ringers, metoclopromide 10mg IV and will have 5g of 0.075% capsaicin cream applied to their abdomen. Participants will indicate the severity of their symptoms immediately prior to administration of metoclopromide, at time 0 and every 30 minutes for a total of 120 minutes after administration of the first medications (or discharge) using a 10 cm visual analogue scale (VAS)11,12. The scale will be provided in English or Spanish as appropriate. If at the 90-minute time mark the patient does not report improvement of their symptoms, odansetron 8mg IV will be administered.
  Interventions: Drug: Capsaicin Topical Cream; Drug: Metoclopramide; Drug: Ondansetron; Drug: Lactated Ringers, Intravenous
- Placebo group (Placebo Comparator): Participants will receive IV fluid bolus of 1000cc of lactated ringers, metoclopromide 10mg IV and will have 5g of placebo cream applied to their abdomen. Participants will indicate the severity of their symptoms immediately prior to administration of metoclopromide, at time 0 and every 30 minutes for a total of 120 minutes after administration of the first medications (or discharge) using a 10 cm visual analogue scale (VAS). The scale will be provided in English or Spanish as appropriate. If at the 90-minute time mark the patient does not report improvement of their symptoms, odansetron 8mg IV will be administered.
  Interventions: Drug: Metoclopramide; Drug: Ondansetron; Drug: Lactated Ringers, Intravenous

INTERVENTIONS:
Drug: Capsaicin Topical Cream — 5g 0.075% applied once
  Arms: Intervention group
Drug: Metoclopramide — 10mg IV once
  Other Names: Reglan
Drug: Ondansetron — 8mg IV once if needed
  Other Names: Zofran
Drug: Lactated Ringers, Intravenous — 1000cc once

SUMMARY:
Between fifty and eighty percent of pregnant women experience nausea and vomiting in pregnancy making it one of the most common medical complications of pregnancy. Hyperemesis gravidarum is an extreme form of nausea and vomiting of pregnancy and results in evidence of acute starvation (i.e. large ketonuria), and weight loss (>5% of a woman's pre-pregnancy weight). Hyperemesis gravidarum is also surprisingly common. In fact, it is the second leading cause of preterm hospitalization during pregnancy, second only preterm labor. Hospitalization is often required because hyperemesis is frequently refractory to common anti-nausea medications. However, capsaicin cream, a potent TRPV1 agonist, commonly used to relieve muscular and neuropathic pain, may be able to reduce the symptoms of nausea and emesis in patients with nausea and vomiting of pregnancy. Smaller studies have demonstrated capsaicin to be both safe and effective when used to treat intraoperative nausea during cesarean delivery. To begin to address whether capsaicin cream could be used to reduce preterm admissions and shorten emergency room visits for hyperemesis, this study will randomize women presenting to the emergency room for nausea and vomiting to treatment with capsaicin cream as an adjunctive medication or routine care. The project will investigate the impact of capsaicin cream on hospital length of stay as well as representation for additional treatment. If effective, capsaicin cream has the potential not only to reduce emergency room visits, hospital admissions and overall health care costs, but also to drastically improve patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the first trimester (0-14 weeks gestation)
* Presenting to the emergency room at Women & Infants Hospital in Rhode Island with a chief complaint of nausea and vomiting
* English or Spanish speaking
* Have not taken an anti-emetic such as Reglan or Zofran within the 6 hours prior to presentation

Exclusion Criteria:

* Allergy to Reglan, capsaicin or Zofran
* Another identifiable source for nausea and vomiting (i.e. gastritis, COVID, diabetic ketoacidosis)
* Molar pregnancies,
* Patients with a history of gastroparesis
* Patients with a history of preexisting diabetes mellitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Murphy, MD, Principal Investigator — Women and Infants Hospital
Locations (1):
- Women and Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bleehen SS. Pigmented basal cell epithelioma. Light and electron microscopic studies on tumours and cell cultures. Br J Dermatol. 1975 Oct;93(4):361-70. doi: 10.1111/j.1365-2133.1975.tb06509.x. PMID 1201188
- [Background] Piwko C, Koren G, Babashov V, Vicente C, Einarson TR. Economic burden of nausea and vomiting of pregnancy in the USA. J Popul Ther Clin Pharmacol. 2013;20(2):e149-60. Epub 2013 Jul 10. PMID 23913638
- [Background] Gazmararian JA, Petersen R, Jamieson DJ, Schild L, Adams MM, Deshpande AD, Franks AL. Hospitalizations during pregnancy among managed care enrollees. Obstet Gynecol. 2002 Jul;100(1):94-100. doi: 10.1016/s0029-7844(02)02024-0. PMID 12100809
- [Background] Richards JR, Lapoint JM, Burillo-Putze G. Cannabinoid hyperemesis syndrome: potential mechanisms for the benefit of capsaicin and hot water hydrotherapy in treatment. Clin Toxicol (Phila). 2018 Jan;56(1):15-24. doi: 10.1080/15563650.2017.1349910. Epub 2017 Jul 21. PMID 28730896
- [Background] Dean DJ, Sabagha N, Rose K, Weiss A, France J, Asmar T, Rammal JA, Beyer M, Bussa R, Ross J, Chaudhry K, Smoot T, Wilson K, Miller J. A Pilot Trial of Topical Capsaicin Cream for Treatment of Cannabinoid Hyperemesis Syndrome. Acad Emerg Med. 2020 Nov;27(11):1166-1172. doi: 10.1111/acem.14062. Epub 2020 Jul 20. PMID 32569429
- [Background] Yuan LJ, Qin Y, Wang L, Zeng Y, Chang H, Wang J, Wang B, Wan J, Chen SH, Zhang QY, Zhu JD, Zhou Y, Mi MT. Capsaicin-containing chili improved postprandial hyperglycemia, hyperinsulinemia, and fasting lipid disorders in women with gestational diabetes mellitus and lowered the incidence of large-for-gestational-age newborns. Clin Nutr. 2016 Apr;35(2):388-393. doi: 10.1016/j.clnu.2015.02.011. Epub 2015 Mar 2. PMID 25771490
- [Background] Yosipovitch G, Mengesha Y, Facliaru D, David M. Topical capsaicin for the treatment of acute lipodermatosclerosis and lobular panniculitis. J Dermatolog Treat. 2005 Aug;16(3):178-80. doi: 10.1080/09546630510041079. PMID 16096187
- [Background] Boogaerts JG, Vanacker E, Seidel L, Albert A, Bardiau FM. Assessment of postoperative nausea using a visual analogue scale. Acta Anaesthesiol Scand. 2000 Apr;44(4):470-4. doi: 10.1034/j.1399-6576.2000.440420.x. PMID 10757584
- [Derived] Murphy LM, Whelan AR, Griffin LB, Hamel MS. A pilot randomized control trial of topical capsaicin as adjunctive therapy for nausea and vomiting of pregnancy. Am J Obstet Gynecol MFM. 2023 Jul;5(7):100997. doi: 10.1016/j.ajogmf.2023.100997. Epub 2023 Jun 2. PMID 37271593

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Placebo Group
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Placebo Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [20 to 30] | 28 [25 to 33] | 26.5 [23 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Parity [Median (Inter-Quartile Range); unit: deliveries] | 1 [0 to 2] | 1 [0 to 2] | 1 [0 to 2]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 23.5 [22 to 27.5] | 22.9 [20.2 to 24.9] | 23.4 [20.95 to 24.88]
Gestational age [Median (Inter-Quartile Range); unit: days] | 68 [54 to 74] | 52 [46 to 66] | 59.5 [49 to 72]

OUTCOME MEASURES:

1. Primary Outcome: Time to Symptom Control
Description: Time to perceived symptom control as measured by time elapsed between metoclopramide administration and patient request for discharge.
Time Frame: 180 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Intervention Group | Placebo Group
Number analyzed (Participants) | 15 | 15
minutes | 72 [56 to 86] | 87 [69 to 111]

2. Secondary Outcome: Number of Antiemetics Needed for Symptom Control
Time Frame: 180 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Placebo Group
Number analyzed (Participants) | 15 | 15
Participants
  1 additional antiemetic | 2 | 4
  2 additional antiemetics | 1 | 1
  3 additional antiemetics | 1 | 0
  4 additional antiemetics | 0 | 0
  0 additional antiemetics | 11 | 10

ADVERSE EVENTS:
Time Frame: Data collected over length of emergency room visit an average of 1.5 hours per participant
Description: Patients self reported side effects
Arm/Group | Intervention Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 10/15 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=15) | Placebo Group (N=15)
Skin irritation (Skin and subcutaneous tissue disorders) | 10 (10) | 0 (0) — Skin irritation including burning and itching

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT05098067/Prot_SAP_ICF_000.pdf